CLINICAL TRIAL: NCT02867735
Title: A Randomized, Single-masked, Sham-control, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of Intravitreal LKA651 in Patients With Macular Edema From Diabetic Macular Edema (DME), Neovascular Age-related Macular Degeneration (AMD), or Retinal Vein Occlusions (RVO)
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of Intravitreal LKA651 in Patients With Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLKA651X2104
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Macular Edema; Diabetic Macular Edema; Neovascular Age-related Macular Degeneration; Retinal Vein Occlusions
Keywords: Macular Edema; Diabetic Macular Edema (DME); Neovascular age-related Macular Degeneration(AMD); Retinal Vein Occlusions (RVO)
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LKA651 (Experimental)
  Interventions: Drug: LKA651
- Sham Comparator (Sham Comparator)
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: LKA651 — Interventional
  Arms: LKA651
Other: Sham Comparator
  Arms: Sham Comparator

SUMMARY:
To evaluate the safety and tolerability of LKA651 in patients with macular edema from diabetic macular edema (DME), neovascular age-related macular degeneration (AMD), or retinal vein occlusions (RVO)

ELIGIBILITY:
Inclusion Criteria:

-Patients with macular edema with center involvement in at least one eye, including those with focal or diffuse DME, neovascular AMD, or RVO

The ETDRS letter score in the study eye must be 60 letters or worse (approximate Snellen equivalent of 20/63)

Vital signs as specified within the protocol

Exclusion Criteria:

-Proliferative diabetic retinopathy in the study eye, with the exception of tufts of neovascularization less than one disc area with no vitreous hemorrhage

Patient, with type 1 or type 2 diabetes who have a hemoglobin A1C > or = 12% at screening

other ocular conditions as specified in the protocol

systemic conditions as specified in the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Number Of participants with Adverse Events as a measure of Safety and Tolerability | Day 1 through study completion
  To evaluate the safety and tolerability of LKA651 by reviewing any adverse events after medical or ophthalmic examinations that are possibly or probably related to study drug.

SECONDARY OUTCOMES:
Pharmacokinetics of Single Dose of LKA651 - Area Under the Curve (AUC) | Plasma samples were collected at Days 1,2,5,8,15,29,43,57,71,85
  To evaluate the serum pharmacokinetic profile of LKA651 Measured by AUC(0-last) - Area under the plasma concentration time curve from time zero to the last quantifiable concentration-time point.
Pharmacokinetics of Single Dose of LKA651 - Cmax | Plasma samples were collected at Days 1,2,5,8,15,29,43,57,71,85
  To evaluate the serum pharmacokinetic profile of LKA651 Measured by Cmax - The maximum plasma concentration of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (5):
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Augusta, Georgia
- Novartis Investigative Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com